CLINICAL TRIAL: NCT01457638
Title: Inferior Turbinate Surgery in Rhinoseptoplasty: a Randomized Clinical Trial With Quality of Life and Acoustic Rhinometry Outcomes
Brief Title: Inferior Turbinate Surgery in Rhinoseptoplasty: a Randomized Clinical Trial With Quality of Life Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1004-20
Record Dates: First submitted 2011-10-17; First posted 2011-10-24 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Nasal Obstruction; Rhinoplasty; Rhinoseptoplasty; Turbinate Surgery; Quality of Life
Keywords: nasal obstruction; rhinoplasty; turbinate surgery; quality of life; acoustic rhinometry
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- No inferior turbinate surgery (Sham Comparator): During rhinoseptoplasty there is no intervention on inferior turbinates
  Interventions: Procedure: No iInferior turbinate surgery
- Inferior Turbinate surgery (Experimental): During rhinoseptoplasty, inferior turbinate submucosal cauterization is performed.
  Interventions: Procedure: Inferior turbinate surgery

INTERVENTIONS:
Procedure: Inferior turbinate surgery — During rhinoseptoplasty inferior turbinate submucosal cauterization is performed.
  Arms: Inferior Turbinate surgery
Procedure: No iInferior turbinate surgery — During rhinoseptoplasty no intervention is done in inferior turbinates
  Arms: No inferior turbinate surgery

SUMMARY:
The purpose of this study is to determine whether inferior turbinate surgery during rhinoseptoplasty is effective in improving quality of life and acoustic rhinometry outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Older than 15 years old;
* Nasal obstruction and nasal aesthetics complaints;

Exclusion Criteria:

* Previous septoplasty, turbinates intervention and/or rhinoplasty;
* Association of other surgical procedures in the same surgical time, as functional endoscopic sinus surgery, blepharoplasty, mentoplasty or otoplasty;
* Inferior turbinate hypertrophy as the isolated cause of nasal obstruction (no septum deviation or internal valve collapse)

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Nasal Obstructive Symptoms Evaluation Scale | 3 months postop
  Specif instrument for evaluation of quality of life related to nasal obstruction

SECONDARY OUTCOMES:
Acoustic Rhinometry | 3 months post-op
World Health Organization Quality of Life (WHOQOL) | 3 months postop
  quality of life instrument
Rhinoplasty Outcomes Evaluation | 3 months postop
  quality of life for rhinoplasty patients
Allergic Conjunctivitis | 3 months postop
  At 90 posoperative day patients were asked if they had allergic conjunctivitis for more than one hour a day on most days, or not.
Nasal Rhinorrea | 3 months postop
  At 90 posoperative day patients were asked if they had nasal rhinorrea for more than one hour a day on most days, or not.
Nasal pruritis | 3 months posopt
  At 90 posoperative day patients were asked if they had nasal pruritis for more than one hour a day on most days, or not.
Nasal Sneeze | 3 months postop
  At 90 posoperative day patients were asked if they had nasal sneeze for more than one hour a day on most days, or not.
Topic nasal corticosteroid | 3 months
  At 90 posoperative day patients were asked if they were using topic nasal corticosteroid or not.
Oral antihistamine | 3 months
  At 90 posoperative day patients were asked if they had used oral antihistamine in the past 30 days or not

CONTACTS AND LOCATIONS:
Overall Officials: Michelle L Wolff, Principal Investigator — Hospital de Clinicas de Porto Alegre/ Universidade Federal do Rio Grande do Sul; Carisi A Polanczyck, PhD, Study Chair — Federal University of Rio Grande do Sul; José E Dolci, PhD, Study Chair — Faculdade de Ciências Médicas da Santa Casa de São Paulo
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Garcia JPT, Moura BH, Rodrigues VH, Vivan MA, Azevedo SM, Dolci JEL, Migliavacca R, Lavinsky-Wolff M. Inferior Turbinate Reduction during Rhinoplasty: Is There Any Effect on Rhinitis Symptoms? Int Arch Otorhinolaryngol. 2021 Aug 5;26(1):e111-e118. doi: 10.1055/s-0041-1726046. eCollection 2022 Jan. PMID 35096167
- [Derived] Lavinsky-Wolff M, Camargo HL Jr, Barone CR, Rabaioli L, Wolff FH, Dolci JE, Polanczyk CA. Effect of turbinate surgery in rhinoseptoplasty on quality-of-life and acoustic rhinometry outcomes: a randomized clinical trial. Laryngoscope. 2013 Jan;123(1):82-9. doi: 10.1002/lary.23628. Epub 2012 Oct 15. PMID 23070968